CLINICAL TRIAL: NCT00642473
Title: A Phase II Trial Assessing Metronidazol Actavis 1% Topical Cream in the Prevention and Treatment of Erlotinib Associated Rash
Brief Title: A Study of Metronidazole Cream in the Prevention and Treatment of Tarceva (Erlotinib)-Associated Rash
Acronym: MATER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21308; 2007-002895-32 (EudraCT Number)
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (2):
- Prevention (Erlotinib + Metronidazole Actavis) (Experimental): Participants will receive erlotinib orally daily. Metronidazole actavis treatment will be initiated at the same day as the start of erlotinib. Metronidazole actavis 1% topical cream will be applied on the right side of the face and chest twice daily for 4 weeks. Left side of the face and chest will be treated according to local standard procedures (ie, with non-active moisturizing cream).
  Interventions: Drug: Erlotinib; Drug: Metronidazole Actavis; Other: Non-active Moisturizing Cream
- Treatment (Erlotinib + Metronidazole Actavis) (Experimental): Participants will receive erlotinib orally daily. Metronidazole actavis treatment will be initiated when participants develop rash. Metronidazole actavis 1% topical cream will be applied on the right side of the face and chest twice daily for 4 weeks. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream).
  Interventions: Drug: Erlotinib; Drug: Metronidazole Actavis; Other: Non-active Moisturizing Cream

INTERVENTIONS:
Drug: Erlotinib — Participants will receive erlotinib 150 milligrams (mg) orally daily for 4 weeks.
  Other Names: Tarceva
Drug: Metronidazole Actavis — Metronidazole actavis 1% topical cream will be applied on the face and chest twice daily for 4 weeks.
Other: Non-active Moisturizing Cream — Left side of the face and chest will be treated according to local standard procedures (ie, with non-active moisturizing cream).

SUMMARY:
This study will evaluate the efficacy and safety of metronidazole actavis 1 percent (%) topical cream in the prevention and treatment of rash associated with Tarceva treatment, in participants with non-small cell lung cancer. The first cohort of participants enrolled in the study will be treated twice daily with metronidazole cream on the right side of the face and upper thorax, the same day as they start treatment with Tarceva (150 mg orally daily). The corresponding body parts on the left side will be treated according to local standard procedures (ie, with non-active moisturizing cream). The second cohort of Tarceva-treated participants will only receive twice daily treatment with metronidazole cream if and when they develop rash. In both cohorts, efficacy will be evaluated at Week 2 and Week 4. The anticipated time on metronidazole treatment is less than (<) 3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer
* eligible to start treatment with erlotinib

Exclusion Criteria:

* hypersensitivity to metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Sweden (6):
  - Gothenburg
  - Lund
  - Malmo
  - Stockholm
  - Umeå
  - Vaxjo

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevention (Erlotinib + Metronidazole Actavis): Participants received erlotinib 150 milligrams (mg) orally daily. Metronidazole actavis treatment was initiated the same day as the start of erlotinib. Metronidazole actavis 1% topical cream was applied on the right side of the face and chest twice daily for 4 weeks to evaluate whether it was effective in the prevention of erlotinib associated rash. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream).
- Treatment (Erlotinib + Metronidazole Actavis): Participants received erlotinib 150 mg orally daily. Metronidazole actavis treatment was initiated when participants developed rash. Metronidazole actavis 1% topical cream was applied on the right side of the face and chest twice daily for 4 weeks to evaluate whether it was effective in the treatment of erlotinib associated rash. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream).
Period: Overall Study
Arm/Group | Prevention (Erlotinib + Metronidazole Actavis) | Treatment (Erlotinib + Metronidazole Actavis)
Started | 18 | 16
Completed | 14 | 5
Not Completed | 4 | 11
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Progression or death | 2 | 4
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Prevention (Erlotinib + Metronidazole Actavis): Participants received erlotinib 150 mg orally daily. Metronidazole actavis treatment was initiated the same day as the start of erlotinib. Metronidazole actavis 1% topical cream was applied on the right side of the face and chest twice daily for 4 weeks to evaluate whether it was effective in the prevention of erlotinib associated rash. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream).
- Total: Total of all reporting groups
Arm/Group | Prevention (Erlotinib + Metronidazole Actavis) | Treatment (Erlotinib + Metronidazole Actavis) | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.8) | 70 (13.1) | 69 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Erlotinib Associated Rash Stratified by Severity Grade at Week 2
Description: Severity of the rash was evaluated semi-quantitatively using the scale of Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0). Grade 0: no rash; Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening or disabling; Grade 5: Death related to rash. Same participant may be counted in more than one reported categories.
Time Frame: After 2 weeks of metronidazole treatment
Population: All enrolled participants. Here, number of participants analyzed = participants who were evaluable for this outcome in respective arms.
Measure: Number; unit: percentage of participants
Groups:
- Left Side - Prevention (Erlotinib + Standard Procedures): Participants received erlotinib 150 mg orally daily for 4 weeks. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream) to evaluate whether it was effective in the prevention of erlotinib associated rash .
- Right Side - Prevention (Erlotinib + Metronidazole Actavis): Participants received erlotinib 150 mg orally daily. Metronidazole actavis treatment was initiated when participants developed rash. Metronidazole actavis 1% topical cream was applied on the right side of the face and chest twice daily for 4 weeks to evaluate whether it was effective in the prevention of erlotinib associated rash.
- Left Side - Treatment (Erlotinib + Standard Procedures): Participants received erlotinib 150 mg orally daily for 4 weeks. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream) to evaluate whether it was effective in the treatment of erlotinib associated rash.
- Right Side - Treatment (Erlotinib + Metronidazole Actavis): Participants received erlotinib 150 mg orally daily. Metronidazole actavis treatment was initiated when participants developed rash. Metronidazole actavis 1% topical cream was applied on the right side of the face and chest twice daily for 4 weeks to evaluate whether it was effective in the treatment of erlotinib associated rash.
Arm/Group | Left Side - Prevention (Erlotinib + Standard Procedures) | Right Side - Prevention (Erlotinib + Metronidazole Actavis) | Left Side - Treatment (Erlotinib + Standard Procedures) | Right Side - Treatment (Erlotinib + Metronidazole Actavis)
Number analyzed (Participants) | 9 | 9 | 6 | 6
percentage of participants
  Facial Rash: Grade 0 (n=9,9,6,6) | 11 | 22 | 0 | 33
  Chest Rash: Grade 0 (n=9,9,6,6) | 56 | 56 | 33 | 50
  Facial Rash: Grade 1 (n=9,9,6,6) | 33 | 22 | 50 | 33
  Chest Rash: Grade 1 (n=9,9,6,6) | 33 | 33 | 17 | 17
  Facial Rash: Grade 2 (n=9,9,6,6) | 22 | 33 | 33 | 17
  Chest Rash: Grade 2 (n=9,9,6,6) | 11 | 11 | 33 | 17
  Facial Rash: Grade 3 (n=9,9,6,6) | 33 | 22 | 17 | 17
  Chest Rash: Grade 3 (n=9,9,6,6) | 0 | 0 | 17 | 17
  Facial Rash: Grade 4 (n=9,9,6,6) | 0 | 0 | 0 | 0
  Chest Rash: Grade 4 (n=9,9,6,6) | 0 | 0 | 0 | 0
  Facial Rash: Grade 5 (n=9,9,6,6) | 0 | 0 | 0 | 0
  Chest Rash: Grade 5 (n=9,9,6,6) | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Erlotinib Associated Rash Stratified by Severity Grade at Week 4
Description: Severity of the rash was evaluated semi-quantitatively using the scale of CTCAE v3.0. Grade 0: no rash; Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening or disabling; Grade 5: Death related to rash. Same participant may be counted in more than one reported categories.
Time Frame: After 4 weeks of metronidazole treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Left Side - Prevention (Erlotinib + Standard Procedures): Participants received erlotinib 150 mg orally daily for 4 weeks. Left side of the face and chest was treated according to local standard procedures (ie, with non-active moisturizing cream) to evaluate whether it was effective in the prevention of erlotinib associated rash.
Arm/Group | Left Side - Prevention (Erlotinib + Standard Procedures) | Right Side - Prevention (Erlotinib + Metronidazole Actavis) | Left Side - Treatment (Erlotinib + Standard Procedures) | Right Side - Treatment (Erlotinib + Metronidazole Actavis)
Number analyzed (Participants) | 8 | 8 | 4 | 4
percentage of participants
  Facial Rash: Grade 0 (n=8,8,4,4) | 13 | 25 | 0 | 25
  Chest Rash: Grade 0 (n=8,8,4,4) | 75 | 63 | 25 | 50
  Facial Rash: Grade 1 (n=8,8,4,4) | 63 | 50 | 50 | 50
  Chest Rash: Grade 1 (n=8,8,4,4) | 0 | 13 | 25 | 25
  Facial Rash: Grade 2 (n=8,8,4,4) | 13 | 25 | 25 | 50
  Chest Rash: Grade 2 (n=8,8,4,4) | 13 | 13 | 25 | 25
  Facial Rash: Grade 3 (n=8,8,4,4) | 0 | 0 | 0 | 0
  Chest Rash: Grade 3 (n=8,8,4,4) | 0 | 13 | 0 | 0
  Facial Rash: Grade 4 (n=8,8,4,4) | 13 | 0 | 0 | 0
  Chest Rash: Grade 4 (n=8,8,4,4) | 13 | 0 | 0 | 0
  Facial Rash: Grade 5 (n=8,8,4,4) | 0 | 0 | 0 | 0
  Chest Rash: Grade 5 (n=8,8,4,4) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 4
Description: Adverse events were not coded using MedDRA or any other standard coding dictionary. Rash was considered an efficacy parameter only and was not considered an adverse event for this study.
Arm/Group | Prevention (Erlotinib + Metronidazole Actavis) | Treatment (Erlotinib + Metronidazole Actavis)
Serious Adverse Events (participants affected / at risk) | 3/18 | 5/16
Other Adverse Events (participants affected / at risk) | 6/18 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Erlotinib + Metronidazole Actavis) (N=18) | Treatment (Erlotinib + Metronidazole Actavis) (N=16)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Falling (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Erlotinib + Metronidazole Actavis) (N=18) | Treatment (Erlotinib + Metronidazole Actavis) (N=16)
Diarrhea (Gastrointestinal disorders) | 4 | 1
Aphthae (Gastrointestinal disorders) | 1 | 0
Pain (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.